CLINICAL TRIAL: NCT06151912
Title: The Effect of Staple Line Reinforcement Procedures on Postoperative Nausea and Vomiting in Sleeve Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: E-16214662-050.01.04-254590-62
Record Dates: First submitted 2023-11-02; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Bariatric Surgical Procedures; Nausea, Postoperative; Vomiting, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Quality of Life

STUDY DESIGN:
Intervention Model Description: Morbidly obese patients will undergo sleeve gastrectomy, starting 3 cm cranial to the pylorus, under the guidance of a 36 F bougie. After gastrectomy, fibrin glue will be applied to the stapler line in one of the groups. In the other group, the staple line will be sutured with 3/0 prolene in an inverted manner.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibrin Glue Group (Experimental): Sleeve gastrectomy will be performed on morbidly obese patients, starting 3 cm cranial to the pylorus, under the guidance of a 36 F bougie. Then, Fibrin Glue (TisseelTM-Baxter, USA) will be applied to the staple line.
  Interventions: Other: Postoperative Nausea and Vomiting scala; Other: Quality of life
- Suture Group (Active Comparator): Sleeve gastrectomy will be performed on morbidly obese patients, starting 3 cm cranial to the pylorus, under the guidance of a 36 F bougie. Then, the stapler line will be sutured with continuous sutures with 3/0 prolene suture, with the stapler line inverted.
  Interventions: Other: Postoperative Nausea and Vomiting scala; Other: Quality of life

INTERVENTIONS:
Other: Postoperative Nausea and Vomiting scala — The Nausea and Vomiting Intensity Scale will be used. Patients will be evaluated with this scale at 1, 6, 24 hours and one month. According to this scale, A total score of ≥50 at any time during the study period will be defined as clinically significant nausea and vomiting.
Other: Quality of life — The EuroQol Group (EQ-5D-5L) questionnaire will assess the quality of life in five domains (mobility, personal care, usual activities, pain and anxiety). A higher score indicates more excellent quality of life impairment. The survey will be administered to patients immediately before surgery and 24 hours and four weeks after surgery to establish baseline values.

SUMMARY:
Obesity is a significant public health problem. The only long-term effective treatment method is surgery. The most common surgical procedure is laparoscopic sleeve gastrectomy (LSG). However, after LSG, complications such as gastroesophageal reflux disease (GERD), insufficient weight loss, stenosis in the remnant stomach, and bleeding or leakage in the staple line (SL) may be encountered. The most severe complications are leakage and bleeding in sleeve gastrectomy, which can lead to many morbidities and mortality. Strengthening the staple line is an important option to prevent these complications. Methods such as fibrin adhesives, bioabsorbable patches and stitching of the stapler line are used to strengthen the stapler line.

Nausea and vomiting, which occur in the postoperative period in 40% of patients who have undergone abdominal surgery and constitute a serious problem, are detected at an even higher rate in patients who have undergone bariatric surgery. Additionally, strengthening the staple line with various methods may increase the incidence of nausea and vomiting after LSG. Although there are studies in the literature investigating whether strengthening the staple line with buttress material or suture in laparoscopic sleeve gastrectomy affects the incidence of postoperative nausea and vomiting, there is no study investigating the effect of strengthening the staple line with fibrin glue on the incidence of postoperative nausea and vomiting.

This prospective study aims to reveal whether there is a difference between strengthening the staple line with fibrin glue or suture in LSG regarding the incidence of postoperative nausea and vomiting and its effects on quality of life.

DETAILED DESCRIPTION:
Bleeding and leaks may occur in the stapler line after sleeve gastrectomy. To prevent these complications, the staple line can be strengthened. More than 60% of bariatric surgeons perform interventions to strengthen the staple line in sleeve gastrectomy.

Two surgeons will perform the operations. One of the surgeons will suture the staple line. The other will apply fibrin glue to the stapler line.

Study: It will be held between June 2023 and June 2024. The same anaesthesia protocol will be applied to all patients during the surgery; All patients will be administered fentanyl 2 mg kg-1, propofol 2.5 mg kg-1 and rocuronium 0.6 mg kg-1 based on lean body weight (LBW) for anaesthesia induction after 3 minutes of preoxygenation. After orotracheal intubation is performed under the guidance of a video laryngoscope and endotracheal intubation is confirmed, 1.0 Minimum alveolar concentration (MAC) value sevoflurane and 1:1 oxygen-air will be used for anaesthesia maintenance. Additional doses of rocuronium were administered if surgically necessary. Ventilation will be applied with a tidal volume of 6-8 ml kg-1 according to the ideal body weight for lung protective ventilation, along with a respiratory frequency at a level to ensure normocapnia (EtCO2 35-45 mmHg). For intraoperative analgesia, remifentanil infusion will be administered at a 0.1-0.3 mcg kg-1 min-1 dose according to ideal body weight. All patients will be given 0.15 mg kg-1 (maximum 16 mg) of ondansetron as an antiemetic. In recovery, sugammadex will be used at a 4-8 mg kg-1 dose to reverse the neuromuscular blockade. For acute postoperative analgesia, 100 mg tramadol, 1000 mg paracetamol and 50 mg dexketoprofen will be administered. No routine postoperative antiemetic medication will be used.

Quality of life index and nausea and vomiting score survey forms will be filled out for patients in the preoperative period, at the 6th, 24th hour and 1st postoperative hour. According to these filled-out forms, the patient's nausea and vomiting scores and quality of life scores will be calculated. Patients included in both groups will be compared to these scores.

This study aims to determine whether there is a difference in strengthening the staple line with fibrin glue or sutures in sleeve gastrectomy regarding the incidence of postoperative nausea and vomiting and its effects on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a body mass index of 40 kg/m2 and above

Exclusion Criteria:

* Patients with hiatal hernia, gastritis or ulcer detected during endoscopy
* Smoker
* Patients who have previously had another bariatric procedure
* Patients who have previously undergone gastrointestinal system surgery
* Patients with any contraindications for bariatric surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting intensity scale (6. hours) | Postoperative 6 hours
  Question 1. Have you vomited or had dry-retching?
  1. No 0 point
  2. Once or twice 2 point
  3. Three or more times 50 points
  Question 2. Have you experienced a feeling of nausea? If yes, has your feeling interfered with being able to get out of bed, walking, eating or drinking?
  1. No 0 point
  2. Sometimes 1 point
  3. Often or most of the time 2 point
  4. All of the time 25 point
  Question 3. Has your nausea been mostly:
  1. Varying ("comes and goes") 1point
  2. Constant 2 point
  Question 4. What was the duration of your feeling of nausea (in hours)?
  …, … (hours). If the answer to Q1=c), score=50 Otherwise, select the highest score of Q1 or Q2, the multiply x Q3 x Q4 Postoperative nausea and vomiting intensity score:
Postoperative nausea and vomiting intensity scale (24. hours) | Postoperative 24 hours
  Question 1. Have you vomited or had dry-retching?
  1. No 0 point
  2. Once or twice 2 point
  3. Three or more times 50 points
  Question 2. Have you experienced a feeling of nausea? If yes, has your feeling interfered with being able to get out of bed, walking, eating or drinking?
  1. No 0 point
  2. Sometimes 1 point
  3. Often or most of the time 2 point
  4. All of the time 25 point
  Question 3. Has your nausea been mostly:
  1. Varying ("comes and goes") 1point
  2. Constant 2 point
  Question 4. What was the duration of your feeling of nausea (in hours)?
  …, … (hours). If answer to Q1=c), score=50 Otherwise, select the highest score of Q1 or Q2, the multiply x Q3 x Q4
  Postoperative nausea and vomiting intensity score:
Postoperative nausea and vomits intensity scale (72. hours) | Postoperative 72 hours
  Question 1. Have you vomited or had dry-retching?
  1. No 0 point
  2. Once or twice 2 point
  3. Three or more times 50 points
  Question 2. Have you experienced a feeling of nausea? If yes, has your feeling interfered with being able to get out of bed, walking, eating or drinking?
  1. No 0 point
  2. Sometimes 1 point
  3. Often or most of the time 2 point
  4. All of the time 25 point
  Question 3. Has your nausea been mostly:
  1. Varying ("comes and goes") 1point
  2. Constant 2 point
  Question 4. What was the duration of your feeling of nausea (in hours)?
  …, … (hours). If answer to Q1=c), score=50 Otherwise, select the highest score of Q1 or Q2, the multiply x Q3 x Q4 Postoperative nausea and vomiting intensity score:
Quality of life (index) | Baseline (Index)
  The EuroQol Group (EQ-5D-5L) questionnaire will be used to evaluate quality of life.
  According to the survey, patients will be evaluated in five areas (mobility, self-care, usual activities, pain, and anxiety).
Quality of life (24. hours) | Postoperative 24 hours
  The EuroQol Group (EQ-5D-5L) questionnaire will be used to evaluate quality of life.
  According to the survey, patients will be evaluated in five areas (mobility, self-care, usual activities, pain, and anxiety).
Quality of life (72. hours) | Postoperative 72 hours
  The EuroQol Group (EQ-5D-5L) questionnaire will be used to evaluate quality of life.
  According to the survey, patients will be evaluated in five areas (mobility, self-care, usual activities, pain, and anxiety).
Quality of life (1. month) | Postoperative 1 month
  The EuroQol Group (EQ-5D-5L) questionnaire will be used to evaluate quality of life.
  According to the survey, patients will be evaluated in five areas (mobility, self-care, usual activities, pain, and anxiety).
Postoperative nausea and vomiting intensity scale (1. month) | Postoperative 1 month
  Question 1. Have you vomited or had dry-retching?
  1. No 0 point
  2. Once or twice 2 point
  3. Three or more times 50 points
  Question 2. Have you experienced a feeling of nausea? If yes, has your feeling interfered with being able to get out of bed, walking, eating or drinking?
  1. No 0 point
  2. Sometimes 1 point
  3. Often or most of the time 2 point
  4. All of the time 25 point
  Question 3. Has your nausea been mostly:
  1. Varying ("comes and goes") 1point
  2. Constant 2 point
  Question 4. What was the duration of your feeling of nausea (in hours)?
  …, … (hours). If answer to Q1=c), score=50 Otherwise, select the highest score of Q1 or Q2, the multiply x Q3 x Q4
  Postoperative nausea and vomiting intensity score:

OTHER OUTCOMES:
Age | 1 day First application
  Years
Body Mass Index (Index) | 1 day First application
  kg/m2
Body mass Index | Postoperative 1 month
  kg/m2

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Adapazarı, Turkey (Türkiye)

REFERENCES:
- [Background] Ruiz-Tovar J, Zubiaga L, Munoz JL, Llavero C. Incidence of postoperative nausea and vomiting after laparoscopic sleeve gastrectomy with staple line reinforcement with oversewing and staple line inversion vs buttressing material: A randomized clinical trial. Int J Surg. 2018 Nov;59:75-79. doi: 10.1016/j.ijsu.2018.09.010. Epub 2018 Oct 3. PMID 30292000
- [Background] Naeem Z, Nie L, Drakos P, Yang J, Gan TJ, Pryor AD, Spaniolas K. The Relationship Between Postoperative Nausea and Vomiting and Early Self-Rated Quality of Life Following Laparoscopic Sleeve Gastrectomy. J Gastrointest Surg. 2021 Aug;25(8):2107-2109. doi: 10.1007/s11605-021-04923-4. Epub 2021 Feb 2. No abstract available. PMID 33528788